CLINICAL TRIAL: NCT01715324
Title: Adjuvant Growth Therapy in in Vitro Fertilization: A Randomized Control Trial
Brief Title: Adjuvant Growth Therapy in in Vitro Fertilization
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Clinique Ovo (Industry)
Collaborators: EMD Serono (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OVO-09-03
Record Dates: First submitted 2012-10-24; First posted 2012-10-26 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2022-01

CONDITIONS: Infertility
Keywords: In vitro fertilization; Antagonist protocol; Growth Hormone
MeSH Terms: conditions — Infertility | interventions — Human Growth Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Growth Hormon (Experimental): The participants randomized in the control group will be prescribed a regular antagonist IVF cycle with dose appropriate stimulation medication and will receive 2.5 mg of Adjuvant Growth Hormon (Saizen) daily via subcutaneous injections, from the beginning of the ovarian reserve stimulation until the day of the ovulation triggering.
  Interventions: Drug: Adjuvant Growth Hormon
- Control (No Intervention): The participants randomized in the control group will be prescribed a regular antagonist IVF cycle with dose appropriate stimulation medication without Adjuvant Growth Hormon (Saizen).

INTERVENTIONS:
Drug: Adjuvant Growth Hormon — The treatment group will receive 2.5 mg of Saizen daily via subcutaneous injections, from the beginning of the ovarian reserve stimulation until the day of the ovulation triggering
  Other Names: Saizen
  Arms: Growth Hormon

SUMMARY:
In an In Vitro Fertilization (IVF) cycle super ovulating drugs (gonadotropins) are usually taken to stimulate the ovaries to produce more than one egg. In Vitro Fertilization protocols are constantly under review in order to improve the recruitment of the follicles, which contain the eggs, whilst minimizing the doses of gonadotrophins required, with the ultimate aim of increasing the live birth rate.

DETAILED DESCRIPTION:
The addition of growth hormone, which is a biological hormone that can be synthetically produced, as a supplement to gonadotrophins in an In Vitro Fertilization cycle has been suggested as a way in which In Vitro Fertilization pregnancy rates may be increased.Growth hormone has been shown, in animal and human studies, to be important in the recruitment of follicles.However, to date, only a limited number of clinical studies have been performed in order to assess whether the addition of growth hormone can improve the probability of pregnancy in women undergoing ovarian stimulation for In Vitro Fertilization. As the total number of patients analysed in these studies was small it has not been possible to determine whether if there is any improvement the outcome of an In Vitro Fertilization cycle when a woman is given growth hormone therapy as a supplement during her treatment.

This goal of this study is to determine the effectiveness of using growth hormone therapy as a supplement to the administration of gonadotropins in an antagonist In Vitro Fertilization protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages of 35 to 42
* Primary or secondary infertility)

  * No previous treatment IVF cycle using the same proposed protocol
* Negative pregnancy test at randomization (urine or blood)

Exclusion Criteria:

* Contraindication to Saizen®
* Simultaneous participation in another clinical trial
* follicle stimulating hormone > 12 IU/L and/or anti-mullerian hormone < 0.5 pg/ml
* Body mass index ≥ 35 kg/m2
* Known risk of gestational diabetes
* Administration of any investigational medication three months prior to study enrolment
* Positive results of screening for either partner for HIV antibodies, Hepatitis B (other than surface antibodies present after vaccination) or Hepatitis C
* Not able to communicate in French or English

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 288 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2021-07 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy rate | 7 weeks
  To determine if the clinical pregnancy rate during the course of one treatment cycle in women receiving Growth Hormone daily in addition to gonadotropin-releasing hormone antagonist protocol is significantly higher than those receiving only gonadotropin-releasing hormone antagonist protocol (control group).

SECONDARY OUTCOMES:
Total dose of gonadotropins | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Number of observed follicles | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Number of mature (Metaphase II) oocytes retrieved | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Oocyte morphology | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Fertilization rate | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Embryo morphology | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Embryo cleavage rate | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Number of embryos available | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Number of supernumerary embryos available for cryopreservation | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Implantation rate | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Miscarriage rate | 40 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Live birth rate | 40 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.
Adverse side effects in women | 7 weeks
  To evaluate the effectiveness of Growth Hormon adjuvant therapy in gonadotropin-releasing hormone antagonist protocol when compared to the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Kadoch, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

REFERENCES:
- [Derived] Mourad A, Jamal W, Hemmings R, Tadevosyan A, Phillips S, Kadoch IJ. Empirical use of growth hormone in IVF is useless: the largest randomized controlled trial. Hum Reprod. 2025 Jan 1;40(1):77-84. doi: 10.1093/humrep/deae251. PMID 39673334
- [Derived] Sood A, Mohiyiddeen G, Ahmad G, Fitzgerald C, Watson A, Mohiyiddeen L. Growth hormone for in vitro fertilisation (IVF). Cochrane Database Syst Rev. 2021 Nov 22;11(11):CD000099. doi: 10.1002/14651858.CD000099.pub4. PMID 34808697